CLINICAL TRIAL: NCT01254630
Title: A Phase III Randomized, Placebo-Controlled, Clinical Trial to Study the Safety and Efficacy of V212 in Adult Patients With Solid Tumor or Hematologic Malignancy
Brief Title: A Study to Evaluate the Safety and Efficacy of Inactivated Varicella-zoster Vaccine (VZV) as a Preventative Treatment for Herpes Zoster (HZ) and HZ-related Complications in Adult Participants With Solid Tumor or Hematologic Malignancy (V212-011)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V212-011; CTRI/2012/05/002673 (Registry Identifier: CTRI); 2010-023156-89 (EudraCT Number); V212-011 (Other: Merck Protocol Number)
Record Dates: First submitted 2010-12-03; First posted 2010-12-06 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Herpes Zoster
Keywords: Herpes zoster; vaccine; herpes-zoster-related complications; immunocompromised; herpes zoster-associated pain; solid tumor malignancy; hematologic malignancy
MeSH Terms: conditions — Herpes Zoster; Hematologic Neoplasms | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- V212-STM (Experimental): Participants with STM receiving chemotherapy randomized to receive V212 vaccine given as a 4-dose regimen administered ~30 days apart.
  Interventions: Biological: V212
- V212-HM (Experimental): Participants with HM randomized to receive V212 vaccine given as a 4-dose regimen administered ~30 days apart.
  Interventions: Biological: V212
- Placebo-STM (Placebo Comparator): Participants with STM receiving chemotherapy randomized to receive placebo to V212 vaccine given as a 4-dose regimen administered ~30 days apart.
  Interventions: Biological: Placebo
- Placebo-HM (Placebo Comparator): Participants with HM randomized to receive placebo to V212 vaccine given as a 4-dose regimen administered ~30 days apart.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: V212 — V212 viral antigen for HZ, 0.5 mL subcutaneous (SC) injection per dose, in a four dose regimen, approximately 30 days apart.
  Other Names: Inactivated Varicella-Zoster (VZV) vaccine
  Arms: V212-HM; V212-STM
Biological: Placebo — Vaccine stabilizer for V212 with no virus antigen, 0.5 mL SC injection per dose, in a four dose regimen, approximately 30 days apart.
  Arms: Placebo-HM; Placebo-STM

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to assess the safety and tolerability of V212 when administered to adults with solid tumor malignancy (STM) receiving chemotherapy and to assess the impact of V212 on the development of herpes zoster (HZ) in adults with STM receiving chemotherapy. The primary hypothesis is that vaccination with V212 will reduce the incidence of HZ compared with placebo in adults with STM (lower bound of the 97.5% {one-sided α=0.0125} confidence interval [CI] for the estimated vaccine efficacy in adults with STM be >25%).

Participants with hematologic malignancy (HM) were also enrolled and were to be originally included in the primary and secondary objectives and analyses. After an interim analysis demonstrated clear evidence of futility of V212 in the HM population, enrollment of this population was stopped and all HM-related objectives and analyses were made exploratory and are not reported in this record.

ELIGIBILITY:
Inclusion criteria:

* Has been diagnosed with an STM or HM and is not likely to undergo hematopoietic cell transplant (HCT) and is either ≥18 years of age and receiving a cytotoxic or immunosuppressive chemotherapy regimen OR is ≥ 50 years of age with a hematologic malignancy that is not in remission, whether on therapy or not
* Life expectancy ≥12 months
* Has prior history of varicella, antibodies to VZV (documented prior to receipt of blood products), or residence in a country with endemic VZV infection for ≥30 years or if participant is <30 years old, attended primary or secondary school in a country with endemic VZV infection
* Is highly unlikely to conceive during the time period starting 2 weeks prior to enrollment through 6 months from last vaccination dose
* Female participants of childbearing potential must have a negative serum or urine pregnancy test

Exclusion criteria:

* History of hypersensitivity reaction to any vaccine component
* Prior history of Herpes Zoster within 1 year of enrollment
* Has received or is expected to receive any varicella or non-study zoster vaccine
* Currently receiving or expected to receive long-term antiviral prophylaxis (>4 weeks duration) with activity against herpes simplex virus (HSV), VZV or cytomegalovirus (CMV)
* Is pregnant or breastfeeding or expecting to conceive within the period of 2 weeks prior to enrollment throughout 6 months from last vaccination dose
* Has received a live virus vaccine or is scheduled to receive a live virus vaccine in the period from 4 weeks prior to Dose 1 through 28 days Postdose 4
* Has received an inactivated vaccine or is scheduled to receive an inactivated vaccine in the period between 7 days prior to and 28 days following Doses 1 through 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5305 (Actual)
Dates: Start 2011-06-24 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Zorger AM, Hirsch C, Baumann M, Feldmann M, Brockelmann PJ, Mellinghoff S, Monsef I, Skoetz N, Kreuzberger N. Vaccines for preventing infections in adults with haematological malignancies. Cochrane Database Syst Rev. 2025 May 21;5(5):CD015530. doi: 10.1002/14651858.CD015530.pub2. PMID 40396505
- [Derived] Hirsch C, Zorger AM, Baumann M, Park YS, Brockelmann PJ, Mellinghoff S, Monsef I, Skoetz N, Kreuzberger N. Vaccines for preventing infections in adults with solid tumours. Cochrane Database Syst Rev. 2025 Apr 16;4(4):CD015551. doi: 10.1002/14651858.CD015551.pub2. PMID 40237463
- [Derived] Boeckh MJ, Arvin AM, Mullane KM, Camacho LH, Winston DJ, Morrison VA, Hurtado K, Durrand Hall J, Pang L, Su SC, Kaplan SS, Annunziato PW, Popmihajlov Z; V212 Protocol 001 Trial Group and V212 Protocol 011 Trial Group. Immunogenicity of Inactivated Varicella Zoster Vaccine in Autologous Hematopoietic Stem Cell Transplant Recipients and Patients With Solid or Hematologic Cancer. Open Forum Infect Dis. 2020 Jun 2;7(7):ofaa172. doi: 10.1093/ofid/ofaa172. eCollection 2020 Jul. PMID 32665955
- [Derived] Mullane KM, Morrison VA, Camacho LH, Arvin A, McNeil SA, Durrand J, Campbell B, Su SC, Chan ISF, Parrino J, Kaplan SS, Popmihajlov Z, Annunziato PW; V212 Protocol 011 Trial Team. Safety and efficacy of inactivated varicella zoster virus vaccine in immunocompromised patients with malignancies: a two-arm, randomised, double-blind, phase 3 trial. Lancet Infect Dis. 2019 Sep;19(9):1001-1012. doi: 10.1016/S1473-3099(19)30310-X. Epub 2019 Aug 6. PMID 31399378

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with a diagnosis of solid tumor malignancy (STM) or hematologic malignancy (HM) were enrolled from 328 sites.
Pre-assignment Details: Out of 5507 screened participants, 5305 were randomized. Twenty randomized participants were not included in analyses: 19 participants from a single site identified to have major Good Clinical Practice compliance issues and 1 participant that was not vaccinated. Thus, a total of 5285 were included in analyses.
Period: Overall Study
Arm/Group | V212-STM | V212-HM | Placebo-STM | Placebo-HM
Started | 1348 | 1288 | 1364 | 1285
Received Vaccination 1 | 1328 | 1277 | 1350 | 1275
Received Vaccination 2 | 1255 | 1217 | 1286 | 1226
Received Vaccination 3 | 1198 | 1178 | 1247 | 1194
Received Vaccination 4 | 1155 | 1145 | 1212 | 1160
Completed | 546 | 0 | 552 | 0
Not Completed | 802 | 1288 | 812 | 1285
Not completed — Adverse Event | 36 | 15 | 40 | 8
Not completed — Death | 461 | 151 | 478 | 139
Not completed — Lost to Follow-up | 80 | 26 | 89 | 32
Not completed — Physician Decision | 24 | 8 | 16 | 7
Not completed — Withdrawal by Subject | 201 | 94 | 188 | 89
Not completed — Study terminated by sponsor | 0 | 994 | 0 | 1010
Not completed — Status not recorded | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants included in study analyses. Twenty randomized participants were not included in baseline analyses: 19 participants from a single site identified to have major Good Clinical Practice compliance issues and 1 participant that was not vaccinated.
Groups:
- Total: Total of all reporting groups
Arm/Group | V212-STM | V212-HM | Placebo-STM | Placebo-HM | Total
Number analyzed (Participants) | 1348 | 1288 | 1364 | 1285 | 5285
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (11.5) | 61.0 (14.9) | 57.7 (11.5) | 61.4 (14.5) | 59.4 (13.3)
Age, Customized [Number; unit: Participants]
  Adults (between 18 and 64 years) | 965 | 705 | 981 | 673 | 3324
  From 65 to 84 years | 379 | 558 | 378 | 589 | 1904
  85 years and over | 4 | 25 | 5 | 23 | 57
Age, Customized [Number; unit: Participants]
  <50 years | 299 | 235 | 320 | 223 | 1077
  ≥50 years | 1049 | 1053 | 1044 | 1062 | 4208
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 867 | 528 | 892 | 523 | 2810
  Male | 481 | 760 | 472 | 762 | 2475
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 17 | 2 | 14 | 2 | 35
  Asian | 55 | 110 | 64 | 94 | 323
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 3 | 2 | 9
  Black or African American | 86 | 41 | 92 | 57 | 276
  White | 1044 | 976 | 1031 | 986 | 4037
  More than one race | 144 | 157 | 159 | 141 | 601
  Unknown or Not Reported | 0 | 0 | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Confirmed Herpes-Zoster
Description: Clinical criteria for suspected HZ cases were the development of a papular or vesicular rash with a dermatomal or generalized distribution, or in the absence of a rash, clinical suspicion of VZV infection with or without the detection of VZV in diagnostic specimens from blood, cerebrospinal fluid, lung, liver, or other organ. All suspected cases of HZ were subjected to adjudication by the Clinical Adjudication Committee (CAC). Case confirmation was based on skin lesion polymerase chain reaction, if available, or by adjudication of the clinical case description by the CAC, conducted according to the CAC Standard Operations Procedure.
Time Frame: Up to approximately 5 years
Population: This analysis was based on the Modified Intent-to-Treat (MITT) population. The MITT population for this outcome measure included all randomized participants in the STM population who received at least one dose of vaccination. This endpoint was exploratory for the HM population, therefore that group was not included in this analysis.
Measure: Number (95% Confidence Interval); unit: Number of cases per 1000 person years
Arm/Group | V212-STM | Placebo-STM
Number analyzed (Participants) | 1328 | 1350
Number of cases per 1000 person years | 6.737 [4.222 to 10.200] | 18.457 [14.118 to 23.709]
Statistical Analysis 1: Comparison: V212-STM vs Placebo-STM; Vaccine efficacy was calculated as 1 minus the hazard ratio of HZ in the V212 group versus the placebo group. The success criterion for vaccine efficacy required that the lower bound of the 97.5% Confidence Interval (CI) be >0.25; Test type: Superiority; Vaccine Efficacy = 0.636, 97.5% CI 2-sided [0.364 to 0.791] — Point estimate and 97.5% CI of vaccine efficacy (primary endpoint) were obtained from a Cox proportional hazards regression model, adjusting for age (<50 versus ≥50 years of age)

2. Primary Outcome: Percentage of Participants With One or More Serious Adverse Events
Description: An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. A serious adverse event (SAE) is an AE that results in death, is life threatening, results in a persistent or significant disability or incapacity, results in or prolongs an existing hospitalization, is a congenital anomaly or birth defect, is a cancer, is an overdose, or is another important medical event.
Time Frame: Up to 28 days after vaccination 4 (up to approximately 118 days)
Population: The analysis population included all participants who received ≥1 dose of vaccination or placebo and had safety follow-up. Three participants in the STM population were cross-treated, these participants were excluded from the safety analyses. This endpoint was exploratory for the HM population, therefore that group was not included in this analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | V212-STM | Placebo-STM
Number analyzed (Participants) | 1322 | 1346
percentage of participants | 22.5 [20.3 to 24.9] | 21.0 [18.9 to 23.3]
Statistical Analysis 1: Comparison: V212-STM vs Placebo-STM; Test type: Other; Risk Difference (RD) = 1.4, 95% CI 2-sided [-1.8 to 4.5]

3. Secondary Outcome: Incidence of Moderate to Severe Herpes-Zoster-Associated Pain
Description: Moderate to severe HZ-associated pain was defined as 2 or more occurrences of a score of 3 or greater (0-to-10 scale, where 0 is no pain and 10 is pain as bad as you can imagine) on the Zoster Brief Pain Inventory (ZBPI) at any time from HZ onset through the end of the 6 month HZ-follow-up period.
Time Frame: Up to 6 months after onset of HZ (up to approximately 5 years)
Population: This analysis was based on the MITT population. The MITT population for this outcome measure included all randomized participants in the STM population who received at least one dose of vaccination. This endpoint was exploratory for the HM population, therefore that group was not included in this analysis.
Measure: Number (95% Confidence Interval); unit: Number of cases per 1000 person years
Arm/Group | V212-STM | Placebo-STM
Number analyzed (Participants) | 1328 | 1350
Number of cases per 1000 person years | 2.144 [0.862 to 4.417] | 9.380 [6.373 to 13.314]
Statistical Analysis 1: Comparison: V212-STM vs Placebo-STM; Vaccine efficacy was calculated as 1 minus the hazard ratio of HZ in the V212 group versus the placebo group. The success criterion for vaccine efficacy required that the lower bound of the 95% CI be >0.25; Test type: Other; Vaccine Efficacy = 0.771, 95% CI 2-sided [0.480 to 0.899] — Point estimate and 95% CI of vaccine efficacy were obtained from a Cox proportional hazards regression model, adjusting for age (<50 versus ≥50 years of age)

4. Secondary Outcome: Incidence of Herpes-Zoster Complications
Description: The composite efficacy endpoint of the incidence of HZ complications was defined as the occurrence of any of the following during the study: hospitalization or prolongation of hospitalization due to HZ, disseminated HZ (including disseminated HZ rash or VZV viremia), visceral HZ, ophthalmic HZ, neurological impairment due to HZ, or administration of intravenous acyclovir therapy for treatment of HZ.
Time Frame: Up to 6 months after onset of HZ (up to approximately 5 years)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Number of cases per 1000 person years
Arm/Group | V212-STM | Placebo-STM
Number analyzed (Participants) | 1328 | 1350
Number of cases per 1000 person years | 0.306 [0.008 to 1.706] | 2.421 [1.045 to 4.770]
Statistical Analysis 1: Comparison: V212-STM vs Placebo-STM; [analysis description as in outcome 3, analysis 1]; Test type: Other; Vaccine Efficacy = 0.874, 95% CI 2-sided [-0.005 to 0.984] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Incidence of Postherpetic Neuralgia
Description: Postherpetic Neuralgia (PHN) was defined as pain in the area of the HZ rash with pain in the last 24 hours scored as 3 or greater (on a 0 to 10 scale, where 0 is no pain and 10 is pain as bad as you can imagine) on the ZBPI that persists or appears greater than or equal to 90 days after HZ rash onset.
Time Frame: Up to 6 months after onset of HZ (up to approximately 5 years)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Number of cases per 1000 person years
Arm/Group | V212-STM | Placebo-STM
Number analyzed (Participants) | 1328 | 1350
Number of cases per 1000 person years | 0.306 [0.008 to 1.706] | 1.210 [0.330 to 3.099]
Statistical Analysis 1: Comparison: V212-STM vs Placebo-STM; [analysis description as in outcome 3, analysis 1]; Test type: Other; Vaccine Efficacy = 0.746, 95% CI 2-sided [-1.275 to 0.972] — [estimate comment as in outcome 3, analysis 1]

6. Other Pre Specified Outcome: Percentage of Participants With Study Medication Withdrawn Due to an Adverse Event
Description: as for outcome 2
Time Frame: Up to 28 days after vaccination 4 (up to approximately 118 days)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | V212-STM | Placebo-STM
Number analyzed (Participants) | 1322 | 1346
percentage of participants | 2.2 | 1.7
Statistical Analysis 1: Comparison: V212-STM vs Placebo-STM; Test type: Other; Risk Difference (RD) = 0.5, 95% CI 2-sided [-0.6 to 1.6]

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to approximately 5 years after vaccination 1.
Description: The All Subjects as Treated population included all participants who received ≥1 dose of vaccination or placebo and had safety follow-up. Three participants in the STM population were cross-treated, these participants were excluded from the safety analyses.
Arm/Group | V212-STM | V212-HM | Placebo-STM | Placebo-HM
All-Cause Mortality (participants affected / at risk) | 472/1322 | 159/1274 | 488/1346 | 146/1274
Serious Adverse Events (participants affected / at risk) | 794/1322 | 500/1274 | 808/1346 | 507/1274
Other Adverse Events (participants affected / at risk) | 857/1322 | 779/1274 | 759/1346 | 559/1274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V212-STM (N=1322) | V212-HM (N=1274) | Placebo-STM (N=1346) | Placebo-HM (N=1274)
Anaemia (Blood and lymphatic system disorders) | 9 (9) | 16 (19) | 24 (25) | 11 (11)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 21 (23) | 44 (64) | 35 (37) | 35 (43)
Haematotoxicity (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4) | 5 (5) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 7 (8) | 5 (5) | 9 (12) | 5 (5)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (6) | 4 (5) | 5 (5) | 4 (4)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 6 (6) | 6 (6) | 5 (5)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aortic valve sclerosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 7 (8) | 9 (12) | 11 (11) | 15 (15)
Atrial flutter (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 8 (8) | 4 (4) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 6 (6) | 3 (3) | 4 (4) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 9 (11) | 11 (12) | 6 (7) | 10 (15)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Cardiomyopathy acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (2)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 4 (4) | 4 (4) | 4 (4)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Pericardial haemorrhage (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular dyssynchrony (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysplastic naevus syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurosensory hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carcinoid syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blindness transient (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cortical visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Necrotising retinitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 3 (3) | 7 (8) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 7 (8) | 1 (1) | 8 (8) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 17 (20) | 1 (1) | 13 (15) | 3 (3)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 5 (5) | 1 (1)
Enteritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 (8) | 6 (6) | 13 (13) | 5 (5)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (3) | 0 (0) | 4 (5) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal fibrosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 12 (16) | 3 (4) | 10 (12) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (3) | 5 (6) | 1 (1)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic insufficiency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 4 (5) | 1 (1) | 2 (2) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Salivary gland calculus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 21 (43) | 4 (4) | 12 (17) | 5 (7)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (11) | 2 (4) | 13 (16) | 3 (3)
Adverse drug reaction (General disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 6 (6) | 4 (4) | 12 (13) | 8 (9)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Death (General disorders) | 31 (31) | 13 (13) | 17 (17) | 7 (7)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 5 (5) | 1 (1) | 3 (3) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Granuloma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Medical device pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Nodule (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Organ failure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Polyserositis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 11 (11) | 5 (5) | 15 (15) | 13 (14)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ulcer haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular stent thrombosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visceral pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biloma (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 4 (5) | 0 (0) | 7 (8) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemobilia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 4 (4) | 1 (1) | 2 (2) | 2 (2)
Graft versus host disease (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hypersensitivity (Immune system disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abscess soft tissue (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anal abscess (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2) | 6 (6) | 3 (3)
Appendicitis perforated (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Bacillus bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 6 (6) | 3 (3)
Bacterial sepsis (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Bacterial tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 10 (10) | 6 (6) | 6 (6)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 4 (4)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 12 (19) | 13 (18) | 19 (21) | 13 (14)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Citrobacter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clostridial sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 9 (9) | 2 (2) | 5 (6) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 2 (2) | 1 (1) | 4 (4) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 7 (7) | 4 (5) | 10 (10) | 2 (2)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Disseminated cryptococcosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (5) | 2 (4)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 4 (4) | 2 (2) | 2 (2) | 4 (4)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal oesophagitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 6 (6) | 5 (5) | 5 (5) | 4 (5)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Genital herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemophilus bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatosplenic candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 4 (4)
Herpes zoster disseminated (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Herpes zoster oticus (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Infected fistula (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected seroma (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 4 (4) | 3 (3) | 6 (7)
Intestinal fistula infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Listeria sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 3 (4)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mediastinitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis cryptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningoencephalitis herpetic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraspinal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleurisy viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 49 (57) | 72 (83) | 49 (53) | 66 (87)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia moraxella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Pneumonia pseudomonal (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Post procedural sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 3 (3) | 0 (0) | 3 (3) | 1 (1)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Psoas abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyomyositis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory moniliasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 28 (32) | 17 (18) | 21 (23) | 21 (22)
Sepsis syndrome (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 6 (6) | 7 (7) | 7 (7) | 10 (10)
Serratia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Serratia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splenic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stenotrophomonas sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Urinary tract infection (Infections and infestations) | 19 (20) | 11 (11) | 24 (24) | 11 (11)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 3 (3) | 2 (5) | 6 (6) | 4 (5)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varicella zoster pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
West Nile viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Wound abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Eschar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 5 (5) | 2 (2)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 2 (2) | 1 (2) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 3 (3) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural discharge (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural fistula (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Radiation necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiation pericarditis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0) | 3 (3)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomal hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urostomy complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CSF test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prothrombin time abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 16 (16) | 2 (2) | 17 (18) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 3 (4) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (3) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1) | 3 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 7 (9) | 6 (6) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 3 (3) | 2 (2)
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture delayed union (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 5 (6) | 4 (4)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Acute monocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5) | 1 (1) | 5 (6)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1) | 3 (3) | 1 (1)
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 0 (0) | 10 (11) | 2 (2)
Adenocarcinoma of salivary gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaplastic large cell lymphoma T- and null-cell types (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaplastic oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angiocentric lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
B precursor type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 9 (9) | 1 (1) | 20 (20)
B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
B-cell lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
B-cell unclassifiable lymphoma low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (12) | 7 (7) | 9 (10) | 11 (11)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0) | 3 (3) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 94 (98) | 2 (2) | 86 (89) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 27 (27) | 0 (0) | 40 (40) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 12 (12) | 0 (0)
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 8 (8) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 54 (56) | 1 (1) | 62 (67)
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5) | 0 (0) | 7 (7)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clear cell sarcoma of soft tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 55 (61) | 0 (0) | 63 (71) | 3 (3)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 33 (35) | 0 (0) | 24 (27) | 0 (0)
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10) | 0 (0) | 8 (8) | 0 (0)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0) | 5 (5) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 6 (6) | 0 (0) | 4 (4)
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0) | 7 (7) | 0 (0)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ependymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epiglottic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ewing's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ewing's sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Extranodal marginal zone B-cell lymphoma (MALT type) recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fallopian tube cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (13) | 0 (0) | 11 (11) | 2 (2)
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 0 (0) | 8 (8) | 0 (0)
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 11 (12) | 0 (0) | 7 (9)
Hodgkin's disease lymphocyte depletion type stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hodgkin's disease mixed cellularity recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hodgkin's disease nodular sclerosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hodgkin's disease nodular sclerosis recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hodgkin's disease recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1) | 9 (10) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratinising squamous cell carcinoma of nasopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large granular lymphocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Laryngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Light chain disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Liposarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1) | 5 (5) | 1 (1)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4) | 0 (0) | 2 (2) | 0 (0)
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1) | 5 (5) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 52 (52) | 3 (3) | 47 (51) | 1 (1)
Lung squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4) | 0 (0) | 6 (6)
Lymphoma transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphoplasmacytoid lymphoma/immunocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoplasmacytoid lymphoma/immunocytoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant histiocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 6 (6) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 4 (5) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 4 (5) | 0 (0)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Mantle cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medullary carcinoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucinous adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mycosis fungoides recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 12 (14) | 0 (0) | 7 (8)
Myelodysplastic syndrome transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 17 (17) | 0 (0) | 10 (10)
Non-Hodgkin's lymphoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0) | 3 (3)
Non-Hodgkin's lymphoma unspecified histology aggressive (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 (23) | 1 (1) | 18 (23) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 4 (4) | 1 (1)
Non-small cell lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Non-small cell lung cancer stage IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Oesophageal adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 0 (0) | 15 (15) | 0 (0)
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteosarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 27 (30) | 0 (0) | 29 (32) | 1 (1)
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 0 (0) | 3 (4) | 0 (0)
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 0 (0) | 3 (3) | 0 (0)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Ovarian epithelial cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 2 (2) | 17 (18) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 5 (5) | 0 (0)
Pancreatic carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic neuroendocrine tumour metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parathyroid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Peripheral T-cell lymphoma unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peritoneal carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 54 (54) | 0 (0) | 54 (57)
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 8 (8) | 0 (0) | 5 (5)
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Precursor T-lymphoblastic lymphoma/leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Precursor T-lymphoblastic lymphoma/leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (17) | 5 (5) | 10 (14) | 1 (1)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 6 (6) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 5 (5) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25 (34) | 0 (0) | 17 (18) | 1 (1)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 0 (0) | 7 (7) | 0 (0)
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Refractory anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3) | 1 (2) | 0 (0)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Sarcoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) | 0 (0) | 6 (6) | 0 (0)
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 6 (6) | 1 (1) | 5 (5)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 4 (4) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 6 (6) | 4 (5) | 10 (10)
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (6) | 0 (0) | 1 (1)
T-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
T-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Tonsillar neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Uterine leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cerebral microangiopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 8 (8) | 4 (4) | 5 (5) | 3 (3)
Cervical cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic coma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 5 (5) | 1 (1)
Hemiparesis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningeal disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myelitis transverse (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 6 (6) | 2 (3) | 5 (5) | 1 (1)
Senile dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Serotonin syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Simple partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 5 (5) | 1 (1) | 3 (3) | 5 (5)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 5 (5) | 1 (1) | 3 (3)
Vasogenic cerebral oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Device failure (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device leakage (Product Issues) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Stent malfunction (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis in device (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 5 (5) | 0 (0) | 4 (4) | 2 (2)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 12 (12) | 10 (11) | 18 (20) | 10 (10)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 4 (4) | 0 (0) | 4 (4) | 0 (0)
Hypercalcaemic nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micturition disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 5 (5) | 2 (2) | 6 (6) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stag horn calculus (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adnexa uteri mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colpocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital erosion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital lesion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Ovarian disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatic disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatic dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 0 (0) | 3 (4) | 4 (4)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 (14) | 8 (19) | 10 (13) | 7 (10)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 6 (6) | 4 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Paranasal sinus mucosal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 5 (5) | 12 (14) | 10 (10)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 4 (8) | 1 (1)
Pneumonia lipoid (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 5 (5) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 28 (28) | 7 (7) | 19 (20) | 5 (5)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Reactive airways dysfunction syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 8 (8) | 2 (2)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Brow ptosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Arterial thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 14 (14) | 6 (6) | 12 (12) | 7 (7)
Embolism (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hypertensive crisis (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 4 (4) | 4 (4)
Hypovolaemic shock (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V212-STM (N=1322) | V212-HM (N=1274) | Placebo-STM (N=1346) | Placebo-HM (N=1274)
Anaemia (Blood and lymphatic system disorders) | 108 (127) | 51 (61) | 114 (140) | 35 (36)
Neutropenia (Blood and lymphatic system disorders) | 89 (121) | 23 (25) | 92 (125) | 28 (32)
Thrombocytopenia (Blood and lymphatic system disorders) | 67 (88) | 14 (15) | 62 (77) | 24 (28)
Constipation (Gastrointestinal disorders) | 63 (68) | 29 (33) | 81 (97) | 38 (42)
Diarrhoea (Gastrointestinal disorders) | 126 (160) | 70 (83) | 137 (181) | 69 (87)
Nausea (Gastrointestinal disorders) | 163 (222) | 83 (125) | 168 (215) | 79 (105)
Vomiting (Gastrointestinal disorders) | 80 (103) | 35 (51) | 92 (104) | 52 (65)
Fatigue (General disorders) | 136 (159) | 71 (74) | 156 (179) | 66 (72)
Injection site erythema (General disorders) | 371 (865) | 389 (875) | 32 (40) | 68 (89)
Injection site pain (General disorders) | 311 (650) | 373 (741) | 78 (103) | 107 (151)
Injection site pruritus (General disorders) | 68 (106) | 94 (153) | 3 (5) | 7 (7)
Injection site swelling (General disorders) | 291 (663) | 329 (715) | 25 (32) | 51 (63)
Pyrexia (General disorders) | 197 (325) | 180 (291) | 198 (361) | 145 (247)
Nasopharyngitis (Infections and infestations) | 38 (40) | 70 (84) | 58 (63) | 71 (88)
Headache (Nervous system disorders) | 94 (137) | 107 (172) | 114 (192) | 95 (172)
Neuropathy peripheral (Nervous system disorders) | 69 (77) | 13 (13) | 76 (86) | 22 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 66 (71) | 68 (76) | 73 (77) | 65 (71)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-30): https://cdn.clinicaltrials.gov/large-docs/30/NCT01254630/Prot_SAP_000.pdf